CLINICAL TRIAL: NCT03463161
Title: A Phase II Study of Epacadostat + Pembrolizumab in Head and Neck Cancer Patients, Who Failed Prior PD-1/PD-L1 Therapy
Brief Title: Epacadostat and Pembrolizumab in Patients With Head and Neck Cancer That Have Failed Prior Immunotherapy
Acronym: ORKA
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Study stopped early due to investigator conflict of interest.
Sponsor: University of Chicago (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB17-1539
Record Dates: First submitted 2018-03-06; First posted 2018-03-13 (Actual); Results first posted 2020-01-27 (Actual); Last update posted 2020-01-27 (Actual); Status verified 2020-01

CONDITIONS: Head and Neck Squamous Cell Carcinoma; Head and Neck Cancer
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck; Head and Neck Neoplasms | interventions — pembrolizumab; epacadostat

STUDY DESIGN:
Intervention Model Description: Participants will be assigned to one of 2 study groups based on response to prior therapy.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Acquired Resistance Group (Experimental): Participants that have benefited from prior treatment with immunotherapy. Defined as response to prior treatment and/or stable disease lasting at least 5 months and disease worsening seen on most recent imaging.
  Participants will receive Pembrolizumab and Epacadostat.
  Interventions: Drug: Pembrolizumab; Drug: Epacadostat
- Suboptimal Benefit Group (Experimental): Participants that have not benefited from prior treatment with immunotherapy. Defined as stable disease lasting at least 5 months or suboptimal response (11-49% shrinkage of tumors). Disease continues to be stable on most recent imaging.
  Participants will receive Pembrolizumab and Epacadostat.
  Interventions: Drug: Pembrolizumab; Drug: Epacadostat

INTERVENTIONS:
Drug: Pembrolizumab — Pembrolizumab (200mg/kg) given by intravenous infusion every 3 weeks.
  Other Names: Keytruda; MK3476
Drug: Epacadostat — Epacadostat (100mg) taken by mouth twice a day.
  Other Names: INCB024360

SUMMARY:
Study to determine response rate of the combination of pembrolizumab plus epacadostat in patients with head and neck cancers that have received prior immunotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Squamous cell carcinoma of the head and neck (which cannot be surgically removed and not amenable to curative intent therapy)
* Meet criteria for either the Acquired Resistance OR the Suboptimal Benefit Group * Acquired Resistance defined as (i and ii must both be met): i. Prior benefit from anti-PD-1/PD-L1 therapy defined as a) prior response, and/or b) ≥5 months of stable disease (SD). Intervening therapies are allowed.

ii. Progressive Disease (PD) on recent scans

* Suboptimal Benefit is defined as (i and ii must both be met): i. Prolonged stable disease ≥5 months OR Suboptimal response (>10% & <50% shrinkage per RECIST at any evaluation timepoint) ii. Ongoing stable disease on recent scans iii. Last treatment with an anti-PD-1/PD-L1 agent within 6 weeks prior to starting protocol treatment

* Availability of stored tumor tissue OR new tumor biopsy Archival tissue for PD-L1 staining (alternatively a new biopsy (core) at baseline can be used). A minimum of 10 slides is required (unless approval from the PI is obtained)
* Measurable disease
* Known human papillomavirus (HPV) status
* Eastern Cooperative Oncology Group (ECOG) performance status 0 or 1
* Be willing and able to provide written informed consent for the trial.
* Aged 18 years or older
* Demonstrate reasonable organ function
* Women of childbearing potential should have a negative urine or serum pregnancy test
* Women of childbearing potential should be willing to use 2 methods of birth control or be surgically sterile, or abstain from heterosexual activity for the course of the study through 120 days after the last dose of study medication
* Males should agree to use an adequate method of birth control starting with the first dose of study therapy through 120 days after the last dose of study medication

Exclusion Criteria:

* Currently participating and receiving treatment in a research study or has participated in a study of an investigational therapy and received study therapy or used an investigational device within 2 weeks of the first dose of treatment on this study
* Diagnosis of immunodeficiency or is receiving systemic steroid therapy or any other form of immunosuppressive therapy within 7 days prior to the first dose of trial treatment.
* Known history of active TB (Bacillus Tuberculosis)
* Hypersensitivity to pembrolizumab, epacadostat or any of its excipients.
* Has received prior anti-cancer monoclonal antibody (mAb) within 3 weeks prior to study Day 1, or targeted small molecule therapy within 2 weeks prior to study Day 1, or who has not recovered (i.e., ≤ Grade 1 or at baseline) from adverse events due to agents administered more than 4 weeks earlier.
* Has not recovered from prior surgery, chemotherapy or radiation therapy from adverse events due to a previous treatment/ administered agent (i.e., ≤ Grade 1 or return to baseline prior to treatment).

Note: Participants with ≤ Grade 2 neuropathy, any grade hearing loss or tinnitus, or typical side effects from radiotherapy are an exception to this criterion and may qualify for the study.

Note: If subject received major surgery, they must have recovered adequately from the toxicity and/or complications from the intervention prior to starting therapy.

* Has a known additional malignancy that is progressing or requires active treatment. Exceptions include basal cell carcinoma of the skin or squamous cell carcinoma of the skin that has undergone potentially curative therapy or in situ cervical cancer or any tumors that are not likely to influence live expectancy in the subsequent 3 years without active treatment (e.g. low grade prostate cancer in absence of therapy).
* Has known active (=growing) central nervous system (CNS) metastases and/or carcinomatous meningitis. Radiation or resected brain metastasis are acceptable if clinically stable.
* Has active autoimmune disease that has required systemic treatment in the past 2 years (i.e. with use of disease modifying agents, corticosteroids or immunosuppressive drugs). Replacement therapy (eg., thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc.) is not considered a form of systemic treatment.
* Has known history of, or any evidence of active, non-infectious pneumonitis.
* Warfarin use, even if low dose warfarin is not acceptable. However, other anti-coagulants (e.g. aspirin, enoxaparin and heparin derivatives, thrombin inhibitors, etc) are acceptable.
* Has a history or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the trial, interfere with the subject's participation for the full duration of the trial, or is not in the best interest of the subject to participate, in the opinion of the treating investigator.
* Has known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial.
* Is pregnant or breastfeeding, or expecting to conceive or father children within the projected duration of the trial, starting with the pre-screening or screening visit through 120 days after the last dose of trial treatment.
* Has received prior therapy with an IDO inhibiting agent.
* Has a known history of Human Immunodeficiency Virus (HIV) (HIV 1/2 antibodies).
* Has known active Hepatitis B (e.g., HBsAg reactive) or Hepatitis C (e.g., HCV RNA [qualitative] is detected).
* Has received a live vaccine within 30 days of planned start of study therapy.
* Has received MAO-inhibitors (MAOI) or drug which has significant MAOI activity (meperidine, linezolid, methylene blue) within the 21 days before screening.
* History of Serotonin Syndrome after receiving serotonergic drugs.
* History or presence of an abnormal electrocardiogram (ECG) that, in the investigator's opinion, is clinically meaningful. Screening QTc interval > 470 milliseconds is excluded.
* Use of any UGT1A9 inhibitor from screening through follow-up period, including the following: diclofenac, imipramine, ketoconazole, mefenamic acid, and probenecid. See Section 5.11 for more details.
* History of organ transplant that requires use of immunosuppressives.
* Any condition that would jeopardize the safety of the subject or compliance with the Protocol.
* Clinically significant cardiac disease, including unstable angina, acute myocardial infarction within 6 months from Day 1 of study drug administration, New York Heart Association Class III or IV congestive heart failure, and arrhythmia requiring therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2018-03-23 (Actual); Primary Completion 2018-12-04 (Actual); Study Completion 2018-12-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Tanguy Seiwert, MD, Principal Investigator — University of Chicago
Locations (1):
- University of Chicago Medical Center, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Groups:
- Acquired Resistance or Suboptimal Benefit Group: Participants that have or have not benefited from prior treatment with immunotherapy.
Period: Overall Study
Arm/Group | Acquired Resistance or Suboptimal Benefit Group
Started | 2
Completed | 2
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Acquired Resistance or Suboptimal Benefit Group
Number analyzed (Participants) | 2
Age, Continuous [Mean (Full Range); unit: years] | 55.5 [52 to 59]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 2
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 2

OUTCOME MEASURES:

1. Primary Outcome: Response Rate
Description: Rate of clinical disease response (tumor shrinkage) as seen on imaging.
Time Frame: up to 18 months
Measure: Count of Participants; unit: Participants
Arm/Group | Acquired Resistance or Suboptimal Benefit Group
Number analyzed (Participants) | 2
Participants | 0

2. Secondary Outcome: Progression Free Survival
Description: Number of patients that have not had disease worsening across both study groups.
Time Frame: 1 year
Population: Study terminated after two patients were enrolled due to conflict of interest with no further patient follow-up.
Arm/Group | Acquired Resistance or Suboptimal Benefit Group
Number analyzed (Participants) | 0

3. Secondary Outcome: Overall Survival
Description: Number of patients surviving across both study groups.
Time Frame: 1 year
Population: Study terminated after two patients were enrolled due to conflict of interest with no further patient follow-up.
Arm/Group | Acquired Resistance or Suboptimal Benefit Group
Number analyzed (Participants) | 0

4. Secondary Outcome: Side Effects
Description: Number of patients with side effect. Summary of side effects by type is provided in adverse events section below.
Time Frame: 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | Acquired Resistance or Suboptimal Benefit Group
Number analyzed (Participants) | 2
Participants | 2

ADVERSE EVENTS:
Time Frame: 8 months
Arm/Group | Acquired Resistance or Suboptimal Benefit Group
All-Cause Mortality (participants affected / at risk) | 0/2
Serious Adverse Events (participants affected / at risk) | 0/2
Other Adverse Events (participants affected / at risk) | 2/2
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Acquired Resistance or Suboptimal Benefit Group (N=2)
Chest wall pain (Musculoskeletal and connective tissue disorders) | 2
Cough (Respiratory, thoracic and mediastinal disorders) | 1
Constipation (Gastrointestinal disorders) | 1
Neutrophil count decreased (Investigations) | 1
Skin and subcutaneous tissue disorders - Other, specify (Skin and subcutaneous tissue disorders) | 1
GastGastrointestinal disorders - Other, specifyrointestinal disorders - Other, specify (Gastrointestinal disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-04-24): https://cdn.clinicaltrials.gov/large-docs/61/NCT03463161/Prot_SAP_000.pdf